CLINICAL TRIAL: NCT05488314
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of Amivantamab and Capmatinib Combination Therapy in Unresectable Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Amivantamab and Capmatinib Combination Therapy in Unresectable Metastatic Non-small Cell Lung Cancer
Acronym: METalmark
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109260; 61186372PANSC2001 (Other: Janssen Research & Development, LLC); 2022-000485-18 (EudraCT Number); 2023-508256-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib; amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Combination Dose Selection) (Experimental): Participants will receive capmatinib 400 milligrams (mg) orally twice daily from Cycle 1 Day 1, in combination with amivantamab 700 mg intravenous (IV) infusion (for body weight less than 80 kilograms [kg]) or 1050 mg IV infusion (for body weight greater than or equal to 80 kg) once weekly from Cycle 1 Day 1 for 4 weeks and then every 2 weeks from Week 5 (Cycle 2; each cycle of 28 days). Doses will be escalated or de-escalated based on the dose limiting toxicities (DLTs) and the recommended Phase 2 combination dose (RP2CD) will be determined by the study evaluation team (SET).
  Interventions: Drug: Capmatinib; Drug: Amivantamab
- Phase 2 (Dose Expansion) (Experimental): Participants with mesenchymal-epithelial transition (MET) exon 14 skipping mutation who are treatment naïve (Cohort 1A), who have received prior therapy (Cohort 1B), or participants with MET amplification who have received prior therapy (Cohort 1C) will receive capmatinib in combination with amivantamab at the RP2CD determined by the SET in Phase 1.
  Interventions: Drug: Capmatinib; Drug: Amivantamab

INTERVENTIONS:
Drug: Capmatinib — Capmatinib will be administered orally.
Drug: Amivantamab — Amivantamab will be administered as IV infusion.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this study is to identify the recommended Phase 2 combination dose (RP2CD[s]) of the amivantamab and capmatinib combination therapy in participants with non-small cell lung cancer (NSCLC) in Phase 1 (combination dose selection), and to evaluate the antitumor effect of the amivantamab and capmatinib combination therapy in mesenchymal-epithelial transition (MET) exon 14 skipping mutation and MET amplified NSCLC, when administered at the selected RP2CD(s) in Phase 2 (expansion).

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with histologically or cytologically confirmed unresectable Stage IV (metastatic) non-small cell lung cancer (NSCLC) (any histology)
* May have: definitively, locally treated brain metastases that are clinically stable and asymptomatic for greater than (>) 2 weeks and who are off or receiving low-dose corticosteroid treatment (less than or equal to [<=]10 milligrams (mg) prednisone or equivalent) for at least 2 weeks prior to start of study treatment
* May have a prior malignancy (other than the disease under study) the natural history or treatment of which is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A participant of childbearing potential must have a negative serum pregnancy test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

* Medical history of (non-infectious) interstitial lung disease (ILD)/pneumonitis, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Participant has impairment of the gastrointestinal function that could affect absorption of capmatinib or is unable or unwilling to swallow tablets
* Participant has symptomatic central nervous system (CNS) metastases which are neurologically unstable or have required increasing doses of steroids >10 mg prednisone or equivalent within the 2 weeks prior to study entry to manage CNS symptoms
* Participant has uncontrolled tumor-related pain: Symptomatic lesions amenable to palliative radiotherapy (example, bone metastases, or metastases causing nerve impingement) should be treated more than 7 days prior to the administration of the first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse events (AEs) by Severity | Up to 2 years 1 month
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1: Number of Participants with Dose Limiting Toxicities (DLTs) | Cycle 1 (Day 1 through Day 28)
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, hematologic toxicity, pulmonary toxicity, liver enzyme elevation, or treatment delay greater than (>) 28 days due to unresolved toxicity.
Phase 2: Objective Response Rate | Up to 2 years 1 month
  ORR is defined as the percentage of participants who achieve either a confirmed partial response (PR) or complete response (CR), using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Phase 1: Number of Participants with AEs by Severity | Up to 2 years 1 month
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1: Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 2 years 1 month
  Number of participants with abnormalities in clinical laboratory parameters (serum chemistry, hematology, coagulation, serology, and urinalysis) will be reported.
Phase 2: Duration of Response (DoR) | Up to 2 years 1 month
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death from any case, whichever comes first, for participants who have PR or CR.
Phase 2: Disease Control Rate (DCR) | Up to 2 years 1 month
  DCR is defined as the percentage of participants who achieve a PR, CR, or stable disease using RECIST version 1.1.
Phase 2: Progression Free Survival (PFS) | Up to 2 years 1 month
  PFS is defined as the time from first dose date until the date of disease progression or death, whichever comes first, based on investigator assessment using RECIST version 1.1
Phase 2: Overall Survival (OS) | Up to 2 years 1 month
  OS is defined as the time from the date of administration of the first study treatment until the date of death due to any cause.
Phase 2: Time to Subsequent Therapy (TTST) | Up to 2 years 1 month
  TTST is defined as the time from the date of administration of the first study treatment to the start date of the subsequent anticancer therapy following study treatment discontinuation, or death, whichever comes first.
Phase 2 (Cohort 1A): Change from Baseline in Health-related Quality of Life in (HRQoL) as Assessed by European Organization of Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | Baseline up to 2 years 1 month
  EORTC-QLQ-C30 is a self-administered, 30-item questionnaire developed to assess the HRQoL of cancer participants.
Phase 2 (Cohort 1A): HRQoL as Assessed by Non-Small Cell Lung Cancer - Symptom Assessment Questionnaire (NSCLC-SAQ) Scale Score | Up to 2 years 1 month
  NSCLC-SAQ assesses patient-reported symptom severity associated with NSCLC.
Phase 2 (Cohort 1A): HRQoL as Assessed by EuroQol 5-Dimension 5-Level (EQ-5D-5L) Scale Score | Up to 2 years 1 month
  EQ-5D-5L is a self-administered, standardized measure of health status.
Phase 2 (Cohort 1A): HRQoL as Assessed by Patient-reported Outcomes Measurement Information System Short Form Version 2.0 - Physical Function 8c (PROMIS PF 8c) Scale Score | Up to 2 years 1 month
  PROMIS PF 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It assesses activities of daily living, mobility, and global impact of physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (78):
- United States (5):
  - University of Alabama at Birmingham, Comprehensive Cancer Center, Birmingham, Alabama
  - The Oncology Institute of Hope and Innovation, Cerritos, California
  - UCLA, Los Angeles, California
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Virginia Cancer Specialists, Fairfax, Virginia
- Brazil (9):
  - PERSONAL Oncologia de Precisao e Personalizada, Belo Horizonte
  - CIONC Centro Integrado de Oncologia de Curitiba, Curitiba
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- Canada (2):
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
- China (14):
  - Beijing Cancer Hospital, Beijing
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Huizhou Municipal Central Hospital, Huizhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- France (4):
  - Institute Coeur Poumon, Lille
  - CHU de la Timone, Marseille
  - Institut de cancerologie de l'ouest, Saint-Herblain
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
- Germany (6):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Muenster, Münster
- Italy (6):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Ospedale S. Maria Delle Croci, Ravenna
  - Istituto Nazionale Tumori Regina Elena, Rome
- Japan (3):
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Shizuoka Cancer Center, Sunto Gun
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - INSTYTUT GENETYKI I IMMUNOLOGII GENIM Sp z o o, Lublin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - Gachon University Gil Hospital, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Del Mar, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Virgen Macarena, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Turkey (Türkiye) (3):
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Bilkent City Hospital, Çankaya
- United Kingdom (4):
  - University College London Hospitals Nhs Foundation Trust, London
  - Imperial College London and Imperial College Healthcare NHS Trust, London
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency